CLINICAL TRIAL: NCT02079987
Title: An Emergency Department-To-Home Intervention to Improve Quality of Life and Reduce Hospital Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201400005; PCORI-1306-01451 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: ED Patients With Chronic Medical Illnesses
Keywords: Healthcare Coach; Care Transition Intervention; Emergency Department Population; Access to Care

STUDY DESIGN:
Who Masked: Investigator
Masking Description: In the ED, a sealed envelope contains the research participants' study assignment. The envelope remains sealed until completion of informed consent and all baseline study procedures after which unmasking occurs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-to-home care transition intervention (Experimental): The ED-to-home care transition intervention is a coaching intervention. It is a 4-week program that uses an Area Agency on Aging healthcare coach to conduct a home visit and at least 3 follow-up phone calls to help patients develop the skills needed for self-management and to communicate with healthcare providers.
  Interventions: Behavioral: ED-to-home care transition intervention
- Usual Care (Experimental): Patients randomized to usual care will receive verbal and written discharge instructions from the treating ED physician and nurse as is the standard of care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: ED-to-home care transition intervention — The Area Agency on Aging coach's role is to build self-management capabilities for the patient and their caregiver. During each contact, the coach reviews the four components of the Care Transition Intervention: 1: Follow-up Medical Visit. 2: Knowledge of Red Flag Symptoms. 3: Medication Reconciliation. 4: The Personal Health Record (PHR). The coach assists patients use the PHR to document and maintain vital information and to communicate with providers.
  Other Names: Care Transition Intervention
  Arms: ED-to-home care transition intervention
Other: Usual Care — Patients randomized to usual care will receive verbal and written discharge instructions from the treating ED physician and nurse as is the standard of care.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine if assigning older, chronically ill patients a healthcare coach after they leave the Emergency Department (ED) improves their quality of life and reduces the need for hospital-based care.

DETAILED DESCRIPTION:
Investigators will review the ED electronic medical record in real-time to determine ED patients' study eligibility. Older, chronically ill ED patients who are eligible and agree to participate in the study will be randomly assigned to a healthcare coach and Care Transition Intervention or usual, post-ED care.

At the time of enrollment, all subjects will be asked to provide informed consent for study investigators to request Medicare Claims to determine how many ED visits, hospital admissions and doctor office visits the subject had at least 30 days after the index ED visit. All research participants will be asked basic personal information such as age, race, sex, employment and marital status. All subjects will be asked to complete a baseline survey about their quality of life.

If the subject is assigned to the Care Transition Intervention, the healthcare coach will visit the subject at home within 3 days of the ED visit. The coach will talk with the subject about following up with a regular, personal doctor and symptoms that indicate a worsening health condition. The coach will help the subject understand their medicines and help the subject make a personal health record (PHR). The coach will tell the subject about the Area Agency on Aging. If the subject receives usual care, they but will be given the usual discharge instructions from the ED nurse and doctor. If the subject receives the Care Transition Intervention, the coach will also call the subject at least 3 times after the ED visit and review the same items listed above.

All enrolled subjects will be asked to complete a phone survey within 31-60 days of the ED visit. This survey will again ask subjects about their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Medicare beneficiaries
* Community dwelling
* Reside within defined geographical area (to enable home visits)
* Have a working telephone
* Have at least one of the following conditions documented in their electronic medical record: congestive heart failure, chronic obstructive pulmonary disease, coronary artery disease, diabetes, stroke, pneumonia, medical and surgical back conditions (predominantly spinal stenosis), hip fracture, peripheral vascular disease, cardiac arrhythmias, deep venous thrombosis, pulmonary embolism, peptic ulcer disease or hemorrhage

Exclusion Criteria:

* Current diagnosis of psychosis
* Cancer
* Dialysis
* History of organ transplantation
* Dementia without a live-in caregiver, or
* In hospice care
* Reside outside the defined geographical area
* Reside in a skilled nursing or assisted living facility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2014-05-03 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna L Carden, MD, MPH, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health, Gainesville, Florida
  - UF Health, Jacksonville, Florida

REFERENCES:
- [Derived] Schumacher JR, Lutz BJ, Hall AG, Harman JS, Turner K, Brumback BA, Hendry P, Carden DL. Impact of an Emergency Department-to-Home Transitional Care Intervention on Health Service Use in Medicare Beneficiaries: A Mixed Methods Study. Med Care. 2021 Jan;59(1):29-37. doi: 10.1097/MLR.0000000000001452. PMID 33298706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medicare beneficiaries with at least 1 chronic medical condition who presented to the ED during the study period were eligible for study entry. Recruitment dates were 5/3/14-11/30/15. Location types: two hospital EDs in north central Florida
Pre-assignment Details: 1322 subjects signed an informed consent. 221 subjects were not included in the analysis because: 1) they did not have a unique Medicare ID; 2) no claims matching the date of index ED visit (informed consent date); 3) not enrolled in Medicare A & B for 12 months prior to index ED visit and at least 30 days after the ED visit.
Groups:
- ED to Home Care Transition: The ED to home care transition intervention is a 4-week program that uses an Area Agency on Aging coach to conduct a home visit and three follow up phone calls to help patients develop self-management skills and to communicate with healthcare providers.
  ED to home care transition: The Area Agency on Aging coach's role is to build self-management capabilities for the patient and caregiver. During each contact, the coach reviews the four components of the Care Transition Intervention: 1: Follow-up Medical Visit. 2: Knowledge of Red Flag Symptoms. 3: Medication Reconciliation. 4: The Personal Health Record (PHR). The coach assists the patient use the PHR to document and maintain vital information and to communicate with providers.
- Usual Care: Patients randomized to usual care will receive verbal and written discharge instructions from the treating emergency department physician and nurse as is the standard of care.
  Usual Care: Patients randomized to usual care will receive usual, post-ED care.
Period: Overall Study
Arm/Group | ED to Home Care Transition | Usual Care
Started | 557 | 544
Completed | 557 | 544
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants who were continuously enrolled in Medicare parts A & B 12 months prior to admission and had at least 30 days enrollment post index ED visit were included in the analysis.
Groups:
- ED to Home Care Transition: The ED-to-home care transition intervention is a 4-week program that uses an Area Agency on Aging healthcare coach to conduct a home visit and at least 3 follow up phone calls to help patients develop the skills needed for disease self-management and to communicate with their providers.
  ED-to-home care transition: The Area Agency on Aging coach's role is to build self-management capabilities for the patient and caregiver. During each contact, the coach reviews the 4 components of the Care Transition Intervention: 1: Follow-up Medical Visits. 2: Knowledge of disease red flags. 3: Medication reconciliation. 4: The Personal Health Record (PHR). The coach assists patients use the PHR to document and maintain vital information and to communicate with providers.
- Usual Care: Usual Care: Patients randomized to usual care will receive verbal and written discharge instructions from the treating emergency department physician and nurse as is the standard of care.
- Total: Total of all reporting groups
Arm/Group | ED to Home Care Transition | Usual Care | Total
Number analyzed (Participants) | 557 | 544 | 1101
Age, Categorical [Count of Participants; unit: Participants] — Medicare beneficiaries presenting to the ED with at least 1 chronic condition were eligible. 1322 subjects signed an informed consent. 221 subjects were not included in the analysis because: 1) they did not have a unique Medicare ID identified; 2) they had no claims matching the date of index ED visit (informed consent date); 3) they were not enrolled in Medicare A & B for 12 months prior to index ED visit and 30 days after the ED visit.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 118 | 120 | 238
    >=65 years | 439 | 424 | 863
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only participants who were continuously enrolled in Medicare parts A & B 12 months prior to index ED visit and had at least 30 days enrollment post index ED visit were included in the health service use analysis.
  years | 72.5 (8.4) | 72.8 (8.6) | 72.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only participants who met inclusion criteria, were continuously enrolled in Medicare parts A & B 12 months prior to admission and had at least 30 days enrollment post index ED visit were included in the analysis.
  Participants
    Female | 336 | 345 | 681
    Male | 221 | 199 | 420
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants who met inclusion criteria, were continuously enrolled in Medicare parts A & B 12 months prior to admission and had at least 30 days enrollment post index ED visit were included in the analysis.
  Participants
    Hispanic or Latino | 18 | 14 | 32
    Not Hispanic or Latino | 539 | 528 | 1067
    Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants who met inclusion criteria, were continuously enrolled in Medicare parts A & B 12 months prior to admission and had at least 30 days enrollment post index ED visit were included in the analysis.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 259 | 244 | 503
    White | 277 | 277 | 554
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 21 | 23 | 44
Region of Enrollment [Number; unit: participants] — Population: Only participants who were continuously enrolled in Medicare parts A & B 12 months prior to admission and had at least 30 days enrollment post index ED visit were included in the analysis.
  participants
    United States | 557 | 544 | 1101

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Function Between Baseline and 60 Days Post-ED Visit
Description: PROMIS Physical Function instruments measure self-reported capability. Each of 7-items in the physical function instrument used in this study has five response items ranging in value from one to five. Thus, the minimum score for the Physical Function Instrument used is 7 and the maximum score is 35. The raw score is translated to a T-score using PROMIS conversion tables. The T-score rescales the raw score into a standardized score with a mean of 50 and standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Physical Function, a T-score of 60 is one SD better than average. A Physical Function T-score of 40 is one SD worse than average. Change in Physical Function is the difference between baseline and 60 day T-score.
Time Frame: Baseline up to 60 days after index ED Visit
Population: Only study participants who completed the baseline ED and follow-up telephone quality of life surveys were analyzed for this primary outcome measure
Measure: Mean (Standard Error); unit: T-score
Groups:
- ED to Home Care Transition: The ED to home care transition intervention is a 4-week program that uses a Area Agency on Aging coach to conduct a home visit and three follow up phone calls to help patients develop the skills needed for self-management and to communicate with healthcare providers.
  ED to home care transition: The Area Agency on Aging patient advocate's role is to build self-management capabilities for the patient and caregiver. During each contact, the patient advocate reviews the four components of the Care Transition Intervention: 1: Follow-up Medical Visit. 2: Knowledge of Red Flag Symptoms. 3: Medication Reconciliation. 4: The Personal Health Record (PHR). The patient advocate assists the patient use the PHR to document and maintain vital information and to communicate with providers.
Arm/Group | ED to Home Care Transition | Usual Care
Number analyzed (Participants) | 384 | 365
T-score | -1.47 (0.62) | -0.83 (0.67)
Statistical Analysis 1: Comparison: ED to Home Care Transition vs Usual Care; Test type: Superiority; p = 0.49, difference-in-difference analysis; A propensity weighted difference-in-difference approach was taken to account for imbalances in assignment and loss to follow-up

2. Primary Outcome: Change in Anxiety Between Baseline and 60 Days Post-ED Visit
Description: PROMIS Anxiety instruments measure self-reported fear, anxious misery, and hyperarousal. Each of 8-items in the Anxiety Instrument used in this study has five response items ranging in value from one to five. Thus, the minimum score for the Anxiety Instrument used is 8 and the maximum score is 40. The raw score is translated to a T-score using PROMIS conversion tables. The T-score rescales the raw score into a standardized score with a mean of 50 and standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Anxiety, a T-score of 60 is one SD worse than average and an Anxiety T-score of 40 is one SD better than average.
Time Frame: Baseline up to 60 days after index ED Visit
Population: Only participants who completed the baseline ED and follow-up telephone quality of life surveys were analyzed for this primary outcome measure.
Measure: Mean (Standard Error); unit: T-score
Groups:
- Usual Care: Patients randomized to usual care will receive verbal and written discharge instructions from the treating emergency department physician and nurse as is the standard of care.
  Usual Care: Patients randomized to usual care will receive verbal and written discharge instructions from the treating emergency department physician and nurse as is the standard of care.
Arm/Group | ED to Home Care Transition | Usual Care
Number analyzed (Participants) | 384 | 365
T-score | 1.53 (0.76) | 0.21 (0.79)
Statistical Analysis 1: Comparison: ED to Home Care Transition vs Usual Care; Test type: Superiority; p = 0.23, difference-in-difference analysis; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Change in Informational Support Between Baseline and 60 Days Post-ED Visit
Description: PROMIS Informational Support instruments measure perceived availability of helpful information or advice. Each of 5-items in the Informational Support Instrument used in this study has five response items ranging in value from one to five. Thus, the minimum score for the Informational Support Instrument used is 5 and the maximum score is 25. The raw score is translated to a T-score using PROMIS conversion tables. The T-score rescales the raw score into a standardized score with a mean of 50 and standard deviation of 10. A higher PROMIS T-score represents more of the concept being measured. For positively-worded concepts like Informational Support, a T-score of 60 is one SD better than average and a T-score of 40 is one SD worse than average.
Time Frame: Baseline up to 60 days after index ED Visit
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ED to Home Care Transition | Usual Care
Number analyzed (Participants) | 384 | 365
T-score | -1.45 (0.79) | -2.84 (0.91)
Statistical Analysis 1: Comparison: ED to Home Care Transition vs Usual Care; Test type: Superiority; p = 0.25, difference-in-difference analysis — A propensity weighted difference-in-difference approach was taken to account for imbalances in assignment and loss to follow-up

4. Primary Outcome: Number of Participants With Outpatient Visit Claims
Description: This outcome was determined by assessing the number of participants who had one or more Medicare claims for an outpatient visit in the 30 days after the index ED visit.
Time Frame: Within 30 days after index ED visit
Population: Participants with Medicare Claims available at least 30 days after the index ED visit are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ED to Home Care Transition | Usual Care
Number analyzed (Participants) | 557 | 544
Participants | 456 | 417
Statistical Analysis 1: Comparison: ED to Home Care Transition vs Usual Care; Test type: Superiority; p = 0.03, Chi-squared

5. Primary Outcome: Number of Participants With ED Visit Claims
Description: This outcome was determined by assessing the number of participants who had one or more Medicare claims for an ED visit in the 30 days after the index ED visit.
Time Frame: Within 30 days after index ED visit
Population: Participants with Medicare Claims available at least 30 days after the index ED visit are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ED to Home Care Transition | Usual Care
Number analyzed (Participants) | 557 | 544
Participants | 135 | 124
Statistical Analysis 1: Comparison: ED to Home Care Transition vs Usual Care; Test type: Superiority; p = 0.57, Chi-squared

6. Primary Outcome: Number of Participants With In-patient Admission Claims
Description: This outcome was determined by assessing the number of participants who had one or more Medicare claims for a hospitalization in the 30 days after the index ED visit.
Time Frame: Within 30 days after index ED visit
Population: Participants with Medicare Claims available at least 30 days after the index ED visit are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ED to Home Care Transition | Usual Care
Number analyzed (Participants) | 557 | 544
Participants | 87 | 78
Statistical Analysis 1: Comparison: ED to Home Care Transition vs Usual Care; Test type: Superiority; p = 0.87, Chi-squared

ADVERSE EVENTS:
Time Frame: 30 days after the index ED visit.
Description: Definition of adverse event and/or serious adverse event does not differ from the clinical trials.gov definitions. Adverse event data were collected in participants who were enrolled in Medicare parts A & B in the 12 months before and 30 days after the index ED visit.
Groups:
- ED to Home Care Transition: The ED to home care transition intervention is a 4-week program that uses an Area Agency on Aging healthcare coach to conduct a home visit and three follow up phone calls to help patients develop self-management skills and to communicate with healthcare providers.
  ED to home care transition: The Area Agency on Aging coach's role is to build self-management capabilities for the patient and caregiver. During each contact, the coach reviews the four components of the Care Transition Intervention: 1: Follow-up Medical Visit. 2: Knowledge of Red Flag Symptoms. 3: Medication Reconciliation. 4: The Personal Health Record (PHR). The coach assists patient use the PHR to document and maintain vital information and to communicate with providers.
Arm/Group | ED to Home Care Transition | Usual Care
All-Cause Mortality (participants affected / at risk) | 16/557 | 17/544
Serious Adverse Events (participants affected / at risk) | 103/557 | 95/544
Other Adverse Events (participants affected / at risk) | 135/557 | 124/544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ED to Home Care Transition (N=557) | Usual Care (N=544)
All cause mortality + hospitalization (General disorders) | 103 (103) | 95 (95) — 30-day hospitalizations and all cause mortality identified through Medicare Claims.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ED to Home Care Transition (N=557) | Usual Care (N=544)
Return ED Visits (General disorders) | 135 (135) | 124 (124) — Return ED visits within 30 days of index ED visit.

LIMITATIONS AND CAVEATS:
Intervention uptake was approximately 60%. 25% of participants did not respond to the follow-up quality of life survey and quality of life was assessed at only two time points. Outpatient visits were based on billed claims not provider type.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No